CLINICAL TRIAL: NCT00827983
Title: Efficacy and Tolerability of Subcutaneous Progesterone Versus Vaginal Progesterone Gel for Luteal Phase Support in Patients Undergoing In-Vitro Fertilization (IVF)
Brief Title: Subcutaneous Progesterone Versus Vaginal Progesterone Gel for Luteal Phase Support in Patients Undergoing In-Vitro Fertilization (IVF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07EU/Prg06
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2012-12-26 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: In Vitro Fertilization
Keywords: Luteal Phase Support in IVF patients
MeSH Terms: interventions — Progesterone

ARMS (2):
- Progesterone SC (Experimental)
  Interventions: Drug: Progesterone
- Progesterone Vaginal gel (Active Comparator)
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — 25 mg, s.c., once à day
  Arms: Progesterone SC
Drug: Progesterone — 90 mg, vaginally, once à day
  Arms: Progesterone Vaginal gel

SUMMARY:
Prospective, open, randomised, parallel, multicentre, two arm trial comparing a new form of luteal support (S.C.) to an approved comparator (vaginal gel).

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 42 (upon starting COH);
* BMI <30 kg/m2;
* <3 prior ART cycles (IVF, ICSI and related procedures);
* Baseline (day 2-3 of cycling) FSH <15 IU/L and E2 <80 pg/mL;
* Normal uterine cavity as per recent hysterosalpingogram, sonohysterogram or hysteroscopic exam (i.e. no polyp or protruding sub-mucosal fibroid);
* At least 3 retrieved oocytes;
* Patient has given written informed consent.

Exclusion Criteria:

* Intramural uterine fibroids that distort the uterine cavity or polyps >1 cm;
* Stage III or IV endometriosis (endometriomas);
* Hydrosalpinx;
* History of past poor response to COH resulting in canceling ART;
* Use of thawed/donated oocytes;
* Use of thawed/donated embryos;
* Patients affected by pathologies associated with any contraindication of being pregnant;
* Hypersensitivity to study medication;
* Uncontrolled adrenal or thyroid dysfunction;
* Undiagnosed vaginal bleeding;
* History of arterial disease;
* Patients with hepatic impairment;
* Neoplasias (current) or history of neoplasia that may be responsive to progesterone;
* High grade cervical dysplasia;
* Active thrombophlebitis or thromboembolic disorders, or a history of hormone-associated thrombophlebitis or thromboembolic disorders;
* History of recurrent pregnancy loss defined as 3 or more spontaneous miscarriages wherein pregnancy developed to a minimum of a gestational sac on TVUS;
* Participation in a concurrent clinical trial or another trial within the past 2 months;
* Use of concomitant medications that might interfere with the study evaluation;
* Pre-implantation genetic diagnosis/screening.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 683 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Klinik fur Frauenheilkunde und Geburthilfe - Universistät zu Lübeck, Lübeck, Germany
- First Dept. Obstetric and Gynaecology, Semmelweiss University Faculty of Medicine, Budapest, Hungary
- Italy (6):
  - Unità Ospedaliera di Ginecologia e Ostetricia, Ospedale Civico Brunico, Bruneck, Bolzano
  - Istituto Scientifico Universitario San Raffaele, Milan, Milan
  - Università degli Studi di Napoli 'Federico II, Naples, Naples
  - Clinica Mangiagalli, Università di Milano, Milan
  - Azienda Ospedaliero-Sanitaria di Modena, Modena
  - Ospedale Santa Chiara, Università degli studi di Pisa, Pisa
- Switzerland (2):
  - IIRM SA, Sorengo, Canton Ticino
  - Universitätsfrauenklinik Basel, Basel
- United Kingdom (4):
  - Midland Fertility Services, Aldridge, West Midlands
  - St. Bartholomew's Hospital - Center for Reproductive Medicine, London
  - Guy's and St. Thomas' Hospital - Women's Health Department, London
  - The Bridge Center, London

REFERENCES:
- [Derived] Griesinger G, Trevisan S, Cometti B. Endometrial thickness on the day of embryo transfer is a poor predictor of IVF treatment outcome. Hum Reprod Open. 2018 Jan 29;2018(1):hox031. doi: 10.1093/hropen/hox031. eCollection 2018. PMID 30895243
- [Derived] Lockwood G, Griesinger G, Cometti B; 13 European Centers. Subcutaneous progesterone versus vaginal progesterone gel for luteal phase support in in vitro fertilization: a noninferiority randomized controlled study. Fertil Steril. 2014 Jan;101(1):112-119.e3. doi: 10.1016/j.fertnstert.2013.09.010. Epub 2013 Oct 17. PMID 24140033

RESULTS

PARTICIPANT FLOW:
Groups:
- Progesterone SC: Progesterone SC was administered at a daily dosage of 25 mg during a minimum of two weeks (in case of no pregnancy) to a maximum of 10 weeks (in case of pregnancy)
- Progesterone Vaginal Gel: Progesterone Vaginal gel was administered at a daily dosage of 90 mg during a minimum of two weeks (in case of no pregnancy) to a maximum of 10 weeks (in case of pregnancy)
Period: Overall Study
Arm/Group | Progesterone SC | Progesterone Vaginal Gel
Started | 339 (All randomised patients) | 344 (all randomised patients)
Completed | 321 (patients who performed the pregnancy test) | 328 (patients who performed the pregnancy test)
Not Completed | 18 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone SC | Progesterone Vaginal Gel | Total
Number analyzed (Participants) | 339 | 344 | 683
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 339 | 344 | 683
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.8 (4.3) | 33.9 (4.3) | 33.8 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 339 | 344 | 683
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 64 | 64 | 128
  Germany | 24 | 23 | 47
  United Kingdom | 46 | 45 | 91
  Switzerland | 48 | 50 | 98
  Italy | 157 | 162 | 319

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Pregnancy Rate at the End of the Study
Time Frame: 10 weeks after treatment start
Population: ITT population was analysed (i.e. all the randomised patients)
Measure: Number; unit: percentage of randomized patient
Arm/Group | Progesterone SC | Progesterone Vaginal Gel
Number analyzed (Participants) | 339 | 344
percentage of randomized patient | 27.4 [lower limit -9.9%] | 30.5
Statistical Analysis 1: Comparison: Progesterone SC vs Progesterone Vaginal Gel; The non -inferiority hypothesis to be tested for the primary endpoint was that the ongoing pregnancy rate (oPR) in the test group (Pe)was lower than the oPR in the control group (Pc)against the alternative one that the oPR in the test group was equal to or higher than the oPR in the control group. H0 : Pc>= Pe + d(-10%) H1 : Pc< Pe + d(-10%); Test type: Non-Inferiority or Equivalence — The null hypothesis (H0) was tested against the alternative by calculating a two-sided 95% confidence interval for the difference in ongoing pregnancy rates. If the lower bound of the 95% confidence interval was greater than the non-inferiority limit (-10.0%), the null hypothesis was rejected and the test group considered not inferior to the control treatment; p = 0.37, Chi-squared; Difference in pregnancy rates = -3.1, 95% CI 2-sided [-9.9 to 3.7]

2. Secondary Outcome: Delivery Rate and Live Birth Rate
Time Frame: nearly 9 month after treatment start
Population: all the randomised patients were included in the analysis
Measure: Number; unit: percentage of randomised patients
Arm/Group | Progesterone SC | Progesterone Vaginal Gel
Number analyzed (Participants) | 339 | 344
percentage of randomised patients | 26.8 | 29.9
Statistical Analysis 1: Comparison: Progesterone SC vs Progesterone Vaginal Gel; Test type: Superiority or Other; p = 0.37, Chi-squared; Risk Difference (RD) = -3.1, 95% CI 2-sided [-9.87 to 3.68]

3. Secondary Outcome: Implantation Rate
Description: Implantation rate was defined as the mean of the total number of gestational sacs seen divided by the total number of embryos transferred. Values are reported as a percentage.
Time Frame: Four to five weeks after oocytes retrieval
Population: All the patients who had at least one embryo transferred
Measure: Mean (Standard Deviation); unit: percentage of embryos transferred
Arm/Group | Progesterone SC | Progesterone Vaginal Gel
Number analyzed (Participants) | 322 | 331
percentage of embryos transferred | 22.6 (35.0) | 23.1 (33.1)
Statistical Analysis 1: Comparison: Progesterone SC vs Progesterone Vaginal Gel; Test type: Superiority or Other; p = 0.85, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-4.7 to 5.8], Standard Error of Mean 1.33

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 10 weeks of treatment, with a follow-up period of 6 months
Description: All the patients who received at least one dose of the study drug have been included in the adverse event analysis.
Arm/Group | Progesterone SC | Progesterone Vaginal Gel
Serious Adverse Events (participants affected / at risk) | 14/338 | 20/344
Other Adverse Events (participants affected / at risk) | 168/338 | 157/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone SC (N=338) | Progesterone Vaginal Gel (N=344)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 5 (5)
Abortion threatened (Psychiatric disorders) | 3 (3) | 3 (4)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
OHSS (Reproductive system and breast disorders) | 4 (4) | 7 (7)
Ovarian torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone SC (N=338) | Progesterone Vaginal Gel (N=344)
Abdominal distension (Gastrointestinal disorders) | 22 (34) | 26 (35)
Abdominal pain (Gastrointestinal disorders) | 19 (33) | 22 (33)
Nausea (Gastrointestinal disorders) | 17 (26) | 16 (34)
Headache (Nervous system disorders) | 18 (29) | 17 (20)
Breast tenderness (Respiratory, thoracic and mediastinal disorders) | 23 (34) | 21 (22)
Uterine spasm (Reproductive system and breast disorders) | 42 (42) | 60 (60)
vaginal discharge (Reproductive system and breast disorders) | 13 (13) | 60 (60)
vaginal hemorrage (Reproductive system and breast disorders) | 48 (48) | 63 (63)
Vaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 28 (28)
Administration site pain (General disorders) | 168 (168) | 25 (25)
Administration site pruritus (General disorders) | 41 (41) | 33 (33)
administration site swelling (General disorders) | 37 (37) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 26 (26)

LIMITATIONS AND CAVEATS:
no special limitations of the trial were detected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No